CLINICAL TRIAL: NCT06538558
Title: A Phase I, Single-Center, Single-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Pharmacokinetics and Efficacy of Tezampanel for Opioid Withdrawal Syndrome in Treatment-Seeking Patients With Opioid Use Disorder
Brief Title: Study to Assess the Use of Tezampanel for Opioid Withdrawal Syndrome in Treatment-Seeking Patients With Opioid Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Proniras Corporation (Industry)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TZP-OWS-001
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use Disorder
Keywords: opioid; OUD; opioid withdrawal syndrome
MeSH Terms: conditions — Opioid-Related Disorders | interventions — tezampanel

STUDY DESIGN:
Intervention Model Description: Participants will be divided into four dose escalation cohorts. A DSMB safety review will be completed after each cohort (at a minimum) to determine appropriateness of continuing dose escalation.
Who Masked: Participant
Masking Description: Participant remains blinded. Investigator and study sponsor are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): 10 participants will be recruited. The first two participants will receive placebo followed by eight participants who will receive active drug (tezampanel) at the lowest dose level.
  Interventions: Drug: Tezampanel; Drug: Placebo
- Cohort B (Experimental): 10 participants will be recruited. The first two participants will receive placebo followed by eight participants who will receive active drug (tezampanel) at the next highest dose level.
  Interventions: Drug: Tezampanel; Drug: Placebo
- Cohort C (Experimental): 10 participants will be recruited. The first two participants will receive placebo followed by eight participants who will receive active drug (tezampanel) at the next highest dose level.
  Interventions: Drug: Tezampanel; Drug: Placebo
- Cohort D (Experimental): 10 participants will be recruited. The first two participants will receive placebo followed by eight participants who will receive active drug (tezampanel) at the next highest dose level.
  Interventions: Drug: Tezampanel; Drug: Placebo

INTERVENTIONS:
Drug: Tezampanel — Study drug will be given intravenously (mg/kg) at 6 timepoints during study participation
  Other Names: TZP
Drug: Placebo — Placebo will be given intravenously (mg/kg) at 6 timepoints during study participation to a subset of participants in each cohort.
  Other Names: PBO

SUMMARY:
This study is examining the use of Tezampanel (TZP) for treatment of Opioid Withdrawal Syndrome (OWS) in participants with Opioid Use Disorder (OUD). Participants will receive TZP or placebo (PBO) daily on Days 2 - 7 during a 7-day inpatient stay at the research center to determine safety, pharmacokinetic (PK) assessment, and efficacy of TZP for OWS.

DETAILED DESCRIPTION:
This study is a phase I, single-center, single-blind, dose escalation study conducted in four cohorts to characterize the safety, tolerability, PK profile and efficacy of TZP for mitigation of OWS in treatment-seeking participants. Participants must be established in an outpatient treatment program and may be taking either long-acting opioid maintenance medications, methadone/buprenorphine, or short-acting opioids (not yet converted to a long-acting maintenance medication).

ELIGIBILITY:
Inclusion Criteria:

1. Male, female or non-binary, age 18 to 65 years of age at Screening.
2. Diagnosis of Opioid Use Disorder (OUD)
3. Positive Urine Drug Screen (UDS) for opioid(s) at the Screening and Baseline Visits.
4. Recent active/chronic use of short-acting illicit and/or prescribed opioids and/or long-acting Opioid Use Disorder (OUD) maintenance treatments buprenorphine or methadone at the Screening and Baseline Visits.
5. Already engaged and fully assessed in a longitudinal-outpatient treatment program that provides opioid addiction treatment encompassing the full spectrum of opioid maintenance and abstinence (injectable Vivitrol®) treatments, in which the host clinic is prepared and equipped to continue with:

   1. maintenance treatment (methadone or buprenorphine treatment) for study non-completers, or
   2. long-acting injectable naltrexone treatment (Vivitrol®), for completers with next dose delivered approximately 30 days after Study Day 6.
6. Post-menopausal/sterile or agree to use chemical or barrier methods of birth control from time of informed consent through 30 days post last treatment.
7. Stable concomitant medications.
8. Stable concomitant medications for depression, post-traumatic stress disorder, psychotic disorders, and bipolar spectrum disorders if one of the following: SSRI, SNRI, bupropion, MAOI, trazodone, Tricyclic, typical and atypical antipsychotics, lithium, antihistamine, alpha-adrenergic agent, nicotine replacement.
9. Stable concomitant medications: propranolol, prazosin, and clonidine if used for psychiatric reasons, and not to control hypertension at the Baseline Visit and unchanged on Study Day 1.
10. Provide informed consent.
11. Understand and follow Lifestyle Considerations per protocol.

Exclusion Criteria:

1. Clinically at risk or unstable due to:

   1. Active psychosis or mania that is impairing insight, decision-making, perception, or ability to provide informed consent as assessed by the PI or designee during the Screening or Baseline Visits, discussion with the outpatient treatment provider, or at Study Day 1.
   2. Active suicidal ideation or intent as assessed by the PI or designee during the Baseline Visit interview or the C-SSRS on Study Day 1.
   3. Chronic benzodiazepine use, or at significant risk for, or in a state of benzodiazepine withdrawal at the Screening or Baseline Visits, Study Day 1, or in discussion with the outpatient treatment provider.
   4. Alcohol Use Disorder as assessed by the PI or designee with > 14 drinks / week (average of > 2 / day) at the Screening or Baseline Visits or Study Day 1 or in discussion with the outpatient treatment provider.
   5. Seizure disorder; use of anti-convulsant for bipolar disorder, seizure, or chronic pain (including topiramate, gabapentin, carbamazepine, valproic acid) at the Screening or Baseline Visits or Study Day 1.
   6. Cardiac abnormalities including arrythmia, conduction abnormality or baseline QTC prolongation (QTcF > 450 males; 470 females); pacemaker, history of myocardial infarction at the Baseline Visit.
   7. Hypertension, diabetes mellitus, cancer, liver, and/or kidney disease and associated medications at the Screening or Baseline Visits or at Study Day 1.
2. Abnormal safety laboratory results.
3. ALT or AST > 3xs upper limit of normal at Baseline or Study Day 1.
4. Undiagnosed hypertension defined as:

   1. Baseline Visit: BP > 160 / 100 mmHg or heart rate > 120 bpm
   2. Study Day 1: BP ≥ 180 / 120 mmHg or heart rate ≥ 140 bpm that continues after 10 minutes of rest.
5. Temperature > 38.1°C at the Baseline Visit. Temperature > 38.9°C at the Study Day 1.
6. Medications that stimulate the dopamine system pre- or post-synaptically, including L-Dopa, lisdexamfetamine, modafinil, gabapentin, phenobarbital, etc.) at the Screening or Baseline Visits or Study Day 1.
7. Medications for addiction, ADHD, insomnia, or bipolar spectrum disorders involving dopamine system stimulants, benzodiazepines, barbiturates, or mood stabilizers active via GABA or glutamate receptor system (e.g. valproic acid, lamotrigine, carbamazepine, acamprosate, disulfiram) at the Screening or Baseline Visits or Study Day 1.
8. Use of naltrexone or acamprosate (active at opioid or glutamatergic receptors) at the Screening or Baseline Visits or Study Day 1.
9. Significant, active infection (e.g., positive for syphilis, tuberculosis, COVID-19, HBV) at the Baseline Visit.
10. Symptomatic HIV or HCV (detectable viral load) at the Baseline Visit.
11. Pregnancy or breastfeeding at the Screening or Baseline Visits or Study Day 1.
12. Poor venous access at the Baseline Visit or Study Day 1.
13. Participation in a research study involving another investigational drug in the last 3 months at the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate systemic tolerability and safety of intravenous tezampanel administration. | First Dose through Day 10 visit
  Monitoring incidence of dose-limiting toxicities, incidence and severity of treatment emergent adverse events.

SECONDARY OUTCOMES:
To characterize Cmax (maximum concentration) of tezampanel | Day 2 and Day 5 (multiple pre and post dose timepoints)
  Samples will be collected and analyzed at various timepoints per protocol
To characterize Area Under the Curve (AUC) concentration of tezampanel | Day 2 and Day 5 (multiple pre and post dose timepoints)
  Samples will be collected and analyzed at various timepoints per protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No